CLINICAL TRIAL: NCT00163774
Title: Intensive Monitoring of Brain Injured Patients; Icp Monitoring, Transcranial Doppler, Jugular Bulb Oximetry, Brain Oxygenation, Brain Temperature and Microdialysis.
Brief Title: Intensive Monitoring of Brain Injured Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayside Health (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 145/02
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2008-05-19 (Estimated); Status verified 2005-09

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

INTERVENTIONS:
Device: Brain oxygenation and microdialysis catheters

SUMMARY:
Analysis of cerebral blood flow (CBF) and oxygenation using complementary focal and global monitoring techniques will permit the delivery of more informed individualised and 'targeted' therapy on the patient with severe head injury, reduce episodes of secondary brain injury and therefore improve outcomes.

Aims

* To develop a deeper understanding of Cerebral Blood Flow and auto-regulation for TBI patients based on the results of data collected in patients post TBI.
* To establish the basis for further multi modality clinical trials in severely brain injured patients in the future.
* To improve understanding of the various secondary processes that continue to cause neuronal damage after the initial injury, and therefore affect patient outcome.
* To proceed to the second phase of the study, with the introduction of algorithms for treatment.

DETAILED DESCRIPTION:
The ultimate aim of this study is to improve the outcome of patients with severe head injury by reducing secondary brain injury. It is hoped that this will be achieved by improving clinical management through the adoption of Best Practice monitoring measures. The severe head injury population is a disparate clinical group with varying CBF derangements, and complex inter-relationships between the various physiological parameters which are being measured. Common protocol based therapy for all head-injured patients is simplistic and cannot fully accommodate the variations between patients or within an individual brain. We believe that to improve outcome, these individual derangements and patterns have to be identified and the correct therapeutic combinations fashioned on an individual basis. This is not the current practice in Australia. The first phase of this project was completed in March 2004 following the recruitment of ten patients. These patients were intensively monitored and based on the data collected and current international literature we devised a new treatment protocol for patients with severe head injuries. We anticipate that implementation of this new protocol will improve outcome.

We aim to:

* further clarify what the above mentioned relationships between monitoring parameters are, what are the most critical ones and the effect that optimisation of these parameters has on brain swelling, ICP control and on clinical outcome.
* introduce treatment algorithms/protocols to alter the haemodynamic parameters, CPP and ICP and to optimise PbrO2.
* study the patients having decompressive craniectomy using these techniques where possible
* compare patient outcomes to previous outcome studies at the Alfred Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic Brain Injury with a Glascow Coma Score < 9 (ie: severe head injury)
* Traumatic Brain Injury with a Glascow Coma Score > 8 with an intracranial pressure monitor in situ and CTscan evidence of one or more of the following: Cerebral oedema (Marshall grades III & IV), midline shift >5 mm cerebral contusion >3cm, evacuated subdural haematoma
* Enrolled within the first 48 hours after trauma
* Aged 17- 70years

Exclusion Criteria:

* Has had a cardiac arrest at or post the trauma scene
* Pupils are fixed bilaterally and dilated >4mm,GCS=3
* Coagulopathy sufficient to contraindicate surgery
* No chance of survival after consideration of CT and clinical findings
* Patients with lower limb/pelvic trauma excluded from Innercool monitoring only

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2002-11; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kossmann, Professor, Principal Investigator — The Alfred
Locations (1):
- The Alfred Hospital, Melbourne, Victoria, Australia